CLINICAL TRIAL: NCT05057299
Title: Extramedullary Acute Myeloid Leukemia (eAML): Retrospective Single Center Cohort Study, Clinicopathological, Molecular Analysis and Survival Outcomes
Status: Completed | Type: Observational
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Khaled Halahleh, Consultant, Medical Oncologist-BMT consultant, King Hussein Cancer Center
Other Study IDs: 20 KHCC 169
Record Dates: First submitted 2021-09-02; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; leukemia,; myeloid sarcoma; extramedullary disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Sarcoma, Myeloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with extramedullary leukemia(eAML) with myeloid neoplasms
  Interventions: Other: retrospective data analysis

INTERVENTIONS:
Other: retrospective data analysis — chart review, analysis and reporting outcomes

SUMMARY:
Patients with extramedullary leukemia were identified over 10 years (January 2003 to September 2019). Clinicopathological,genetic-molecular features were identified and survival outcomes were studied and analyzed.

DETAILED DESCRIPTION:
We retrospectively collected patients demographics ,including clinicopathological and genetic-molecular parameters in patients with extramedullary leukemia between January 2003 till September 2019 from King Hussein cancer center(KHCC) electronic medical records. All potential prognostic factors were identified and compared with worldwide data published previously. Treatment and survival outcomes were studies and analyzed.

Primary endpoint : Overall survival (OS).

Secondary endpoint :

* Progression Free Survival (PFS).
* incidence of extramedullary leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged ≥18 year and up to 75 years
* Male and females.
* Initially diagnosed and treated with extramedullary leukemia at KHCC and followed till last encounter.
* Patients, who underwent an allogeneic stem cell transplant.
* Period January 2003-September 2019

Exclusion Criteria:

* Pediatric patients <18 year of age
* Patients, who lost their follow up within study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — males and females
Study Population: Patients diagnosed with eAML and treated at medical oncology department of KHCC-lymphoma section between January 2003-september 2019.Patients identified by searching KHCC registry databases, using key terms of myeloid sarcoma, granulocytic sarcoma, chloroma, AML, MDS, MPN, relapse. All clinicopathological and molecular data were collected and cases, that satisfied the WHO criteria for the diagnosis of myeloid sarcoma were included in the study. The clinicopathological data included age, sex, prior diagnoses and treatment, disease location, phenotype using flow cytometry or immunohistochemistry, status of bone marrow disease (prior, concurrent or after diagnosis of eAMl), treatment for eAML and their overall survival.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS), | "4 year, year 4"
  To calculate the median and estimated 4-year overall survival

SECONDARY OUTCOMES:
Progression-Free Survival | "4 year, year 4"
  To calculate the median and estimated 4-year PFS

CONTACTS AND LOCATIONS:
Locations (1):
- King Hussein Cancer Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shallis RM, Wang R, Davidoff A, Ma X, Zeidan AM. Epidemiology of acute myeloid leukemia: Recent progress and enduring challenges. Blood Rev. 2019 Jul;36:70-87. doi: 10.1016/j.blre.2019.04.005. Epub 2019 Apr 29. PMID 31101526
- [Result] Shallis RM, Gale RP, Lazarus HM, Roberts KB, Xu ML, Seropian SE, Gore SD, Podoltsev NA. Myeloid sarcoma, chloroma, or extramedullary acute myeloid leukemia tumor: A tale of misnomers, controversy and the unresolved. Blood Rev. 2021 May;47:100773. doi: 10.1016/j.blre.2020.100773. Epub 2020 Oct 30. PMID 33213985